CLINICAL TRIAL: NCT04684979
Title: A Non-Myeloablative Conditioning Regimen With Peri-Transplant Rituximab and the Transplantation of Hematopoietic Stem Cells From HLA-compatible Related or Unrelated Donors in Patients With B-Cell Lymphoid Malignancies
Brief Title: Transplantation of Hematopoietic Stem Cells From HLA-compatible Donors in Patients With B-Cell Lymphoid Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The landscape of treatment for patients targeted for enrollment has significantly changed since the protocol was written and approved, and the research treatment is no longer the best option for this population.
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KOE-002
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: B-Cell Lymphoid Malignancies; Hematologic Malignancy; Non-Hodgkin Lymphoma
Keywords: Hematologic Malignancies, NHL
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: The study design will be based on a total of 90 patients, 30 recipients of related matched and 60 recipients of mismatched related or unrelated PBSCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HLA-compatible Related Donor (Experimental): This is a phase 2 study to evaluate NMA PBSCT incorporating peri-transplant rituximab and utilizing PBSC to augment graft cell dose in patients with selected B lymphoid malignancies. Salvage chemotherapy will be required as part of transplant eligibility, both to achieve debulking of disease to allow sufficient time for the development of a post-transplant GVL effect, and to contribute to recipient immune suppression and thus facilitate donor engraftment.
  Interventions: Biological: Hematopoietic Stem Cells from HLA-compatible Related
- Unrelated Donor (Experimental): This is a phase 2 study to evaluate NMA PBSCT incorporating peri-transplant rituximab and utilizing PBSC to augment graft cell dose in patients with selected B lymphoid malignancies. Salvage chemotherapy will be required as part of transplant eligibility, both to achieve debulking of disease to allow sufficient time for the development of a post-transplant GVL effect, and to contribute to recipient immune suppression and thus facilitate donor engraftment.
  Interventions: Biological: Hematopoietic Stem Cells from HLA Unrelated

INTERVENTIONS:
Biological: Hematopoietic Stem Cells from HLA-compatible Related — NMA PBSCT (Non-Myeloablative peripheral blood stem cell transplantation) incorporating rituximab and utilizing PBSC (Peripheral blood stem cells) to increase graft cell dose in patients with selected B lymphoid malignancies.
  Arms: HLA-compatible Related Donor
Biological: Hematopoietic Stem Cells from HLA Unrelated — NMA PBSCT (Non-Myeloablative peripheral blood stem cell transplantation) incorporating rituximab and utilizing PBSC (Peripheral blood stem cells) to increase graft cell dose in patients with selected B lymphoid malignancies.
  Arms: Unrelated Donor

SUMMARY:
This research study is being conducted to treat patients with B-cell lymphoid malignancies. These types of cancers include diffuse large cell (DLBCL) non-Hodgkin's lymphoma (NHL), mantle cell NHL, any indolent B cell NHL (such as follicular, small cell or marginal zone NHL), or chronic lymphocytic leukemia (CLL). Patients with these types of lymphomas have been shown to benefit from peripheral blood stem cell transplantation (PBSCT). PBSCT uses healthy blood stem cells from a donor to replace your diseased or damaged bone marrow. Before undergoing PBSCT, you'll receive chemotherapy and/or radiation to destroy your diseased cells and prepare your body for the donor cells. This is called a "conditioning regimen." Non-myeloablative (NMA) conditioning causes minimal cell death. This research study will look at a course of treatment using NMA conditioning regimen including low dose chemotherapy and low dose radiation as well as rituximab and PBSCT from a compatible donor. The primary aim is to obtain a preliminary estimate of the overall and event-free survival 1 year post-transplant after NMA.

DETAILED DESCRIPTION:
This is a phase 2 study of a treatment regimen consisting of a non-myeloablative (NMA) conditioning regimen incorporating low dose chemotherapy and low dose radiation as well as peri-transplant Rituximab and the transplantation of peripheral blood stem cells (PBSC) from an HLA compatible related or unrelated donor in patients with B cell lymphoid malignancies including diffuse large cell (DLBCLC) and mantle cell non-Hodgkin's lymphoma (MCL), indolent B cell NHL, or chronic lymphocytic leukemia (CLL). The study design will be based on a total of 90 patients, 30 recipients of related matched and 60 recipients of mismatched related or unrelated PBSCT.

It is anticipated that the accrual will last 5-6 years. At the conclusion of the study, the safety and a preliminary assessment of efficacy of NMA PBSCT will be determined. The treatment will be declared efficacious if the disease-free survival at 1 year in this patient population is at least 50%.

ELIGIBILITY:
Inclusion Criteria:

* :

  * Patients aged 18-74 years at initial referral with a suitably matched related or unrelated donor who have provided their informed consent to participate in the clinical trial.
  * If post-pubertal, females agree to take hormonal therapy to suppress menses unless a specific contra-indication to estrogen exists

Diagnosis:

* Patients with CD20+ aggressive B cell NHL (DLBCL, large cell transformation of indolent NHL/CLL, or mantle cell) OR CD20+ indolent NHL/CLL. Relapsed disease must be biopsy proven and CD20 positivity must be demonstrated within the 12 months prior to protocol enrollment.

Eligible patients with DLBCL NHL will:

* have relapsed disease following initial therapy but failed to mobilize or had bone marrow involvement and therefore are not suitable for an autologous transplant OR
* have high-intermediate or high-risk second-line age-adjusted International Prognostic Index score and be in 2nd CR/PR following an autologous transplant OR
* have failed an autologous transplant and be in PR or better after salvage chemotherapy.

Eligible patients with transformed indolent NHL/CLL will:

• have CR/PR of the large cell component of their disease after either salvage chemotherapy or an autologous transplant.

Eligible patients with mantle cell NHL will:

* be high-risk such as p53 positivity and be in 1st CR/PR after initial therapy OR
* have relapsed disease following initial therapy and be in 2nd or 3rd CR/PR after salvage chemotherapy.

Eligible patients with indolent B cell NHL (such as, but not limited to, follicular, small cell or marginal zone NHL) or CLL will:

• have 1st or subsequent progression or primary refractory disease (pre-allograft cytoreduction necessary but CR/PR not required).

Pre-allograft Salvage Chemotherapy:

* This can include a single autologous transplant using high dose chemotherapy conditioning if appropriate OR ≥ 2 cycles of intensive combination chemotherapy (e.g. RICE) as appropriate according to diagnosis and prior therapy.
* CLL patients who have received CAMPATH do not have to receive pre-allograft salvage chemotherapy.

Timing of PBSCT:

• Admission for PBSCT must be within 120 days of autologous transplantation OR 80 days of the last cycle of chemotherapy.

Organ Function and Performance Status Criteria:

* Karnofsky score ≥ 70 %
* calculated creatinine clearance ≥ 50 mL/min OR if creatinine ≥ 1.2, a history of renal dysfunction, age > 50 years, prior transplant, and/or a single kidney, the patient must have a measured creatinine clearance (using 24 hour urine collection) ≥ 50 mL/min
* bilirubin < 2.5, AST/ALT ≤ 3 x upper limit of normal (unless benign congenital hyperbilirubinemia)
* pulmonary function (spirometry and corrected DLCO) ≥ 50% normal
* left ventricular ejection fraction ≥ 40%
* albumin ≥ 2.5. Donor HLA-compatible related donors
* Patients who have an HLA-matched or one allele mismatched related donor are eligible for entry on this protocol. This will include a healthy related donor who is genotypically or phenotypically matched at least 9/10 of the A, B, C, DRB1, and DQB1 loci, as tested by high resolution.

HLA-compatible Unrelated donors • Patients who do not have a related HLA-matched donor but have an unrelated donor who is matched at

≥ 9/10 (allele mismatch only) of the A, B, C, DRB1, and DQB1 loci, as tested by high resolution.

Exclusion Criteria:

* Diagnosis: known negativity for CD20 pre-allograft; mantle cell or DLBCL NHL with progressive disease at allograft work-up

  * Prior Therapy: prior allogeneic transplant (prior autologous transplant is acceptable)
  * Cytoreduction and timing of NMA PBSCT: patients unable to complete planned cytoreduction due to therapy complications, or who undergo cytoreduction but are unable to proceed to allografting within the defined time period, are ineligible for allograft on protocol
  * Active and uncontrolled infection at time of transplantation including active infection with Aspergillus or other mold, or HIV infection
  * Patients positive for Hepatitis B or C at risk for viral reactivation.
  * Inadequate performance status/organ function
  * Pregnant or breast feeding
  * Patient or guardian unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up and research tests.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Estimate the overall and event-free survival | 1 year
  The primary aim of this study is to obtain a preliminary estimate of the overall and event-free survival at 1 year after NMA PBSCT with peri-transplant rituximab using an HLA matched or single HLA allele disparate related or unrelated donors

SECONDARY OUTCOMES:
Speed of Recovery Post Allograft | 100 days
  the speed of neutrophil and platelet recovery post allograft
Response to Engraftment | 100 days
  the incidence and speed of donor-derived engraftment
Status of Graft Versus Host Disease | 100 days
  The incidence and severity of acute GVHD(Graft Versus Host Disease) at 100 days
Number of Participants with Graft Versus Host Disease | 1 year
  The incidence and severity of chronic GVHD (Graft Versus Host Disease) at 1 year
Number of Participants with Complications | 100 days
  the incidence of serious infectious complications with their correlation with laboratory measurements of immune recovery
Response Rate to Vaccination | 100 days
  the response to vaccination after PBSCT (Peripheral Blood Stem Cells Transplantation)
Number of Transplant Related Mortality Incidences | 100 and 180 days
  the incidence of Transplant Related Mortality at 100 and 180 days
Number of Relapse or Disease Progression Instances | 1 and 2 years
  the incidence of malignant relapse or disease progression at 1 and 2 years
Number of Overall and Event Free Survival | 2 years
  the probabilities of overall and event-free survival at 2 years after Peripheral Blood Stem Cells Transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Koehne, MD, PhD, Principal Investigator — Miami Cancer Institute at Baptist Health of South Florida
Locations (1):
- Miami Cancer Institute at Baptist Health of South Florida, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Miami Cancer Institute Website — http://baptisthealth.net/cancer-care/home